CLINICAL TRIAL: NCT06512649
Title: Early Recognition and Intervention in Siblings at High-risk for Neurodevelopmental Disorder
Acronym: ERI-SIBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: University of Milano Bicocca (Other); Politecnico di Milano (Other); Catholic University of the Sacred Heart (Other); University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 94-7
Record Dates: First submitted 2024-06-03; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-05

CONDITIONS: Neurodevelopmental Disorders; Autism Spectrum Disorder
MeSH Terms: conditions — Neurodevelopmental Disorders; Autism Spectrum Disorder | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early Intervention Group (Experimental): ASD and typical siblings with Signs of concern
  Interventions: Behavioral: Early intervention
- Clinical Monitoring Group (No Intervention): Typical siblings with no signs of concern Children allocated to this arm will undergo to re-assessment at T1 and T2
- Active monitoring Group (Experimental): ASD siblings, no signs of concern
  Interventions: Behavioral: Active monitoring

INTERVENTIONS:
Behavioral: Early intervention — 90-minute parent-coaching session once a week for 6 months with an expert developmental therapist, supported by a child neuropsychiatrist or psychologist. A parent will always be present and actively involved in the intervention. The intervention is individualized and tailored to each child's needs and identifies with caregivers the ways to embody objectives in daily life.
  Arms: Early Intervention Group
Behavioral: Active monitoring — 90-minute session once a month for 6 months. Sessions will be performed by an expert developmental therapist, supported by a child neuropsychiatrist or psychologist. A parent will always be present and actively involved in the intervention.
  Arms: Active monitoring Group

SUMMARY:
H1The primary goal of this intervention study is to learn if very early parent-mediated intervention in children at risk for neurodevelopmental disorders in the first year of life can be implemented in routine care, positively impacting early sensory-motor and socio-communicative developmental trajectories and reducing the developmental gap in children with signs of concern.

H2: It is here postulated that early intervention with active parental involvement can reduce parental stress, as well as improve parental understanding and responsiveness to the child's communication cues.

H3: An important part of our work will be analysing data about early social and joint attention behaviours in recruited children and comparing them at different time points. The hypothesis is to find early differences between groups at baseline and to detect a change before and after the intervention. For this reason, in our study design, we decided to use technologies to collect data on quantitative measures during play-structured and laboratory sessions to understand changes in developmental trajectories.

H4: Given the potential role of genetic and immunological mechanisms in ASD, one of the study's secondary aims is to investigate the impact of an early intervention programme on epigenetic changes and inflammatory and immune response.

After enrolment and baseline assessments (T0), children will be allocated to the three groups:

* Group 1 - Clinical Monitoring Group (CM): Siblings of TD children subjects with no signs of concern
* Group 2 - Active Monitoring Group (AM): Siblings of ASD children with no signs of concern
* Group 3 - Early Intervention Group (EI): Siblings classified as "with signs of concern" at baseline evaluation.

All children will be re-evaluated after 6 months (T1) and after 12 months (T2).

DETAILED DESCRIPTION:
Researchers will contact interested parents to assess eligibility and provide detailed study information. Parents will provide written consent before completing baseline assessments (T0) and based on the scores at the main outcome measures, children will be assigned to the correct group. Infants with no signs of concern and siblings of TD children will be allocated to Group 1 (CM); infants with no signs of concern (scores at the Griffiths-3 and CSBS-ITC in the normal range) and siblings of ASD children will be allocated to Group 2 (AM); infants with General Quotient score below 85 using Griffiths-3 and/or at least one score above the "concern" cutoff using the CSBS-ITC will be allocated to Group 3 (EI). Families allocated to Groups 2 and 3 will start the intervention within one month from the baseline assessment. Families allocated to Group 1 will perform only the evaluations at different time points. Assessments will be conducted at baseline (T0), which will be when the parents give their consent and within the 8 months of life of the child, after 6 months from the start of the intervention (T1) and after 12 months from the start of the intervention (T2).

Technological assessment of social behaviour and joint attention:

- video recording of ESCP through Kinect Azure camera to collect and analyse quantitative data related to joint attention.

The administration of the ECSP-I will be video-recorded through an Azure Kinect camera to extract automatically gaze orientation and quantitatively assess Joint Attention.

- Eye-tracker acquisitions An experimental Eye-Tracker Screening (ETS) protocol for children will also be developed. Specifically, short videos will be used to measure the children's ability to process familiar/unfamiliar faces and to respond to social stimuli, particularly referential gaze. The children's eye movements will be analysed using the eye-tracker (Tobii Pro Fusion) and extracted using the appropriate software.

At recruitment (T0), anamnestic, sociodemographic data and auxological and clinical parameters at birth will be collected.

Biomolecular assessment Saliva samples will be collected using 3 different kits, respectively for DNA or RNA extraction, and for protein detection, through spongy swabs that are inserted into the baby's mouth, leading the saliva collection non-invasive, simple, fast, and most importantly, painless. Saliva samples will be collected from all the probands (at T0, T1 and T2) and from their siblings and parents at T0 to assess parent-to-child genetic transmission in relation to the risk of ASD. If possible, a sample of approximately 40 mL of blood (from the parents) will be collected.

Biological samples from family quartet will be collected as follow:

1. In all the enrolled children, their older siblings and parents, genetic analysis will be conducted by a Next-Generation Sequencing (NGS) gene-targeted panel approach to analyse genes involved in synaptogenesis and immunogenetic regulation.
2. Epigenetic analysis of the miRNome in saliva collected from all enrolled children at all time-points will be performed by NGS. Epigenetic analysis will allow to define a panel of microRNAs that can differentiate between ASD children and children with typical development.
3. Analysis of inflammatory cytokines and neurotrophic factors using an automated immunoassay system (ELLA, Biotech) will be performed in probands at T0, T1 and T2. Parents will also be characterized for cytokine and lymphocyte subset at T0.

Correlations between clinical parameters and all biological variables (genetic, epigenetic, inflammatory) will be performed to correlate molecular biomarkers with neurodevelopmental changes in follow-up and pre-post intervention.

Sample size

Since the importance of ECSP-I in this project, as behavioural outcome measures as a tool for reaching quantitative data through technology, we calculate the sample size to detect an association between the ECSP-I score and the groups (1, 2 and 3) at each time point. The calculation was performed based on preliminary data (not already published) from the Italian Version of ESCP (ECSP-I). Assuming a standard deviation of 0.56 for the ECSP-I scale and a significance level α= 0. 01, obtained by applying the Bonferroni correction for multiple comparisons, performed in pairs between groups, to the type I error, we obtained a sample size of 14 subjects per group to detect a difference of 0.8 between the means of each group using a 2-tailed Student's t-test for independent samples, with a power of 80%. Assuming a drop-out rate of 10%, the required sample size increases to 16 subjects per group, that is 48 subjects in total.

Statistical analysis

Analysis (using STATA or SPSS 28.00) will follow standard methods for trials using comparisons between the three groups. First, a study of the maturation trajectories of the infants will be carried out, with a description of the pre-post intervention changes in the tests carried out. Secondly, quantitative evaluations of joint attention data and molecular markers will be performed, detected, and described through mean and standard deviation in case of Gaussian distribution of variables, or median and interquartile range in case of non-Gaussian distribution. The normality of distributions will be assessed by applying the Shapiro-Wilk test. For categorical variables, absolute frequencies and percentages will be reported. Genetic analysis of intra-familial allelic inheritance will be conducted by AFBAC (Affected Family-Based Controls) and TDT (Transmission Disequilibrium Test) . The immunological parameters obtained from the groups of ASD children and children with typical development will be analysed using a nonparametric Mann-Whitney test that will allow to identification of specific immunological biomarkers of ASD-associated neuroinflammation. Moreover, clinical parameters will be correlated with immunological biomarkers characteristic of ASD children. Finally, epigenetic analysis will allow us to define a panel of microRNAs that can differentiate between ASD children and children with typical development. Using computer algorithms, the potential targets, pathways, and biological functions deregulated by this group of miRNAs will be analysed. These data will also be analysed concerning the clinical parameters evaluated in the study and both the genetic and inflammatory characterization of the subjects studied.

ELIGIBILITY:
Inclusion Criteria:

* Age at recruitment less than or equal to 8 months.
* Sibling diagnosed with autism spectrum disorder
* Normal neurological examination

Exclusion Criteria:

* Focal neurological signs/symptoms or suspicion of genetic-metabolic disorders
* Genetically determined suspected or known conditions in brother/sister
* Significant familial language barrier

Ages: 6 Months to 8 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Griffiths Scales of Child Development, 3rd Edition (Griffiths-3) | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  Griffiths-3 is the gold standard to provide an overall measure of a child's development (0-6 years); it permits the definition of an individual profile of strengths and needs of the child across five areas: foundations of learning, language and communication, eye and hand coordination, personal-social-emotional, gross motor
  UNIT OF MEASURE: Developmental quotients (range 20-150, normality 85-115)
Communication and Symbolic Behaviour Scales - Infant-Toddler Checklist (CSBS-IT-C) | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  is a tool for developmental screening, designed to measure 7 language predictors in children 6 to 24 months of age. The questions of the checklist may be presented in an interview format with adequate explanations to clarify what is being asked. It takes about 5 to 10 minutes to complete and permits the detection of signs of concern for ASD in infants and toddlers
  UNIT OF MEASURE: weighted score, number: range 3-17; no concern > 7
Early Social Communication Scale (Échelle de la Communication Sociale Précoce, Italian adaptation, ECSP-I) | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  the ECSP-I is a structured assessment designed to provide measures of individual differences in nonverbal communication skills in children from 3 to 30 months of age. The administration requires 15-20 min involving the presentation of approximately 23 standardised situations which provide opportunities for social communication. The ECSP-I demonstrates strong reliability and both construct and discriminant validity
  Unit of measure: number. Optimal and average level (mean, range 1-4).
Satisfaction Survey | T1 (T0 + 6 months)
  Parents of children in Groups 2 and 3 will also be asked to anonymously complete a satisfaction survey (created ad hoc for this project) immediately after the intervention to assess their satisfaction with the services provided. The questionnaire takes 5 minutes to complete.
  unit of measure: likert scale, range 0-5

SECONDARY OUTCOMES:
Vineland Adaptive Behaviour Scales-II - Second Edition (Vineland-II) | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  This assessment measures personal and social adaptation skills in everyday-life. It is applicable to children from birth through 18 years, 11 months. Standardization included national samples of children with and without disabilities.
  The scales yield normative standard scores (M = 100; SD = 15) that indicate level of adaptive functioning
Questionnaire Sensory Profile - Second Edition (SP-2) | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  The SP-2 is a norm-referenced collection of five parent- and teacher-report questionnaires that assess sensory processing in children about everyday sensory events; for this study, the age-appropriate version was used, that is the Toddler Module (from 7 to 35 months); Unit of measure: items are rated on a 5-point Likert scale from 5 (almost always) to 1 (almost never). Point are scored as Standard Deviation through automatized scoring provided by the editor
McArthur-Bates questionnaire, child's first vocabulary (PVB) - gestures and words | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  The PVB assesses major features of communicative development, including words' comprehension and production, use of gesture, and first sentences' comprehension. The PVB/words and gestures form is a checklist filled by the parents'. The questionnaire is validated on an Italian sample, and it allows to calculate quotients related to the different subareas investigated
  Unit of measure: centile according to age (range 5-95) and quotients (number)
Infant Behavior Questionnaire-Revised (IBQ-R) and Early Childhood Behavior Questionnaire (ECBQ) | T0 (recruitment); T2 (T0 + 12 months)
  The IBQ-R (3-12 months) and ECBQ (18-36 months) are parent-report questionnaires for the assessing of temperament in infancy and later childhood; items are rated on a 7-point scale (from 1 that is 1 never to 7 that is always) (Cozzi et al., 2013; Gartstein & Rothbart, 2003)
Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) | T2 (T0 + 12 months)
  The ADOS-2 is a semi structured, standardized assessment of communication social interaction, play/imaginative use of materials and restricted/repetitive patterns of interest to assess the presence of ASD symptoms. The administration involves direct observations using hierarchical manualized procedures and progressive prompts. Every behaviour/symptom is assessed using a likert scale (0-3) and coded on an algorithm based on DSM-5 diagnostic criteria. We will use Toddler Module, for 12 to 30 months-aged children, or the Module 2 if language in sentences is present.
  We will consider the total score (unit of measure number, range 0-28), social affect score (unit of measure number, range 0-20), and restricted and repetitive behaviours score (unit of measure number, range 0-8).
Autism Diagnostic Interview-Revised (ADI-R) | T2 (T0 + 12 months)
  The ADI-R is a semi-structured interview conducted by a trained researcher or psychologist with the child's parents or other caregivers, based on DSM-IV criteria. The ADI-R focuses on the developmental history of the child and on the actual description given by the parents.
  Every behaviour/symptom is assessed using a likert scale (0-3) and coded on an algorithm. We will use algorithms specifically developed for toddlers, that give a clinical cutoff and a rate of risk for ASD.
  unit of measure: number
Parent interactions with children: Checklist of Observations Linked to Outcomes (PICCOLO) | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  this is an observational measure in which a parent-child interaction is video recorded and trained observers code-specific parenting behaviours known to predict children's early social, cognitive, and language development. Specifically, the PICCOLO examines four domains of parenting behaviours, including affection, responsiveness, encouragement, and teaching. The PICCOLO demonstrates strong reliability and both construct and predictive validity.
  Each domain is scored on a 0-2 likert scale.
  Unit of measure: number, range 0-14 for each subscale
Questionnaire Parent Stress Index - Short Form (PSI-SF) | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  It is a questionnaire completed by the parents, composed by thirty-six items are divided into three domains: Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI), and Difficult Child (DC), which combine to form a Total Stress scale.
  UNIT of MEASURE: centiles, number. Range 1-99
Kinect | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  video recording of ESCP through Kinect Azure camera to collect and analyse quantitative data to estimate the gaze orientation.
  * time spent by the child looking at the therapist
  * joint attention lenght, (the time during which the child and the therapist simultaneously focus on the same object or each other).
  Unit of measure: absolute time values (seconds) and a relative measurement in relation to the total session duration (percentage)).
  To date, there are no normative data available in the literature for these specific metrics.
Eye-tracker | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  An experimental Eye-Tracker Screening (ETS) protocol will be implemented using the Tobii Pro Fusion 120Hz to analyze children's eye movement patterns. The indices that will be used include Total Fixation Duration (TFD) and Time to First Fixation (TFF).
  TFD will measure children's general attention to specific areas, such as faces and objects (i.e. target and distractor).TFF will assess children's ability to follow the gaze of the familiar or unfamiliar faces towards the target, thereby verifying their response to referential gaze (i.e., the gaze-following mechanism).
  Both indices, TFD and TFF, will be measured in milliseconds.
Laboratory- genetic analysis | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  genetic analysis will be conducted by a Next-Generation Sequencing (NGS) gene-targeted panel approach to analyse genes involved in synaptogenesis and immunogenetic regulation.
  Gene association will be reported as genotypes and alleles NUMBER and percentages
Laboratory- epigenetic analysis | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  Epigenetic analysis of the miRNome by NGS. Epigenetic analysis will allow to define a panel of microRNAs that can differentiate between ASD children and children with typical development.
  MiRNA concentrations will be reported as COPIES/NANOGRAMS of extracted RNA
Laboratory- inflammatory cytokines and neurotrophic factors | T0 (recruitment), T1 (T0 + 6 months); T2 (T0 + 12 months)
  Analysis of inflammatory cytokines and neurotrophic factors using an automated immunoassay system (ELLA, Biotech).
  Cytokine and neurotrophic factors concentration measured in saliva and plasma samples will be reported as PICOGRAMS/ML.
  Results calculations will be based on standard curves and internal controls provided by commercial kits

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Maria Nascente, Milan, Italy

REFERENCES:
- [Background] Armitano-Lago C, Willoughby D, Kiefer AW. A SWOT Analysis of Portable and Low-Cost Markerless Motion Capture Systems to Assess Lower-Limb Musculoskeletal Kinematics in Sport. Front Sports Act Living. 2022 Jan 25;3:809898. doi: 10.3389/fspor.2021.809898. eCollection 2021. PMID 35146425
- [Background] Baroncelli L, Braschi C, Spolidoro M, Begenisic T, Sale A, Maffei L. Nurturing brain plasticity: impact of environmental enrichment. Cell Death Differ. 2010 Jul;17(7):1092-103. doi: 10.1038/cdd.2009.193. Epub 2009 Dec 18. PMID 20019745
- [Background] Bertram J, Kruger T, Rohling HM, Jelusic A, Mansow-Model S, Schniepp R, Wuehr M, Otte K. Accuracy and repeatability of the Microsoft Azure Kinect for clinical measurement of motor function. PLoS One. 2023 Jan 26;18(1):e0279697. doi: 10.1371/journal.pone.0279697. eCollection 2023. PMID 36701322
- [Background] Colombi C, Chericoni N, Bargagna S, Costanzo V, Devescovi R, Lecciso F, Pierotti C, Prosperi M, Contaldo A. Case report: Preemptive intervention for an infant with early signs of autism spectrum disorder during the first year of life. Front Psychiatry. 2023 May 3;14:1105253. doi: 10.3389/fpsyt.2023.1105253. eCollection 2023. PMID 37205979
- [Background] Di Giovanni D, Enea R, Di Micco V, Benvenuto A, Curatolo P, Emberti Gialloreti L. Using Machine Learning to Explore Shared Genetic Pathways and Possible Endophenotypes in Autism Spectrum Disorder. Genes (Basel). 2023 Jan 25;14(2):313. doi: 10.3390/genes14020313. PMID 36833240
- [Background] Elsabbagh M, Bedford R, Senju A, Charman T, Pickles A, Johnson MH; BASIS Team. What you see is what you get: contextual modulation of face scanning in typical and atypical development. Soc Cogn Affect Neurosci. 2014 Apr;9(4):538-43. doi: 10.1093/scan/nst012. Epub 2013 Feb 5. PMID 23386743
- [Background] Green J, Charman T, Pickles A, Wan MW, Elsabbagh M, Slonims V, Taylor C, McNally J, Booth R, Gliga T, Jones EJ, Harrop C, Bedford R, Johnson MH; BASIS team. Parent-mediated intervention versus no intervention for infants at high risk of autism: a parallel, single-blind, randomised trial. Lancet Psychiatry. 2015 Feb;2(2):133-40. doi: 10.1016/S2215-0366(14)00091-1. Epub 2015 Jan 28. PMID 26359749
- [Background] Green J, Pickles A, Pasco G, Bedford R, Wan MW, Elsabbagh M, Slonims V, Gliga T, Jones E, Cheung C, Charman T, Johnson M; British Autism Study of Infant Siblings (BASIS) Team. Randomised trial of a parent-mediated intervention for infants at high risk for autism: longitudinal outcomes to age 3 years. J Child Psychol Psychiatry. 2017 Dec;58(12):1330-1340. doi: 10.1111/jcpp.12728. Epub 2017 Apr 10. PMID 28393350
- [Background] Guzzetta A, Baldini S, Bancale A, Baroncelli L, Ciucci F, Ghirri P, Putignano E, Sale A, Viegi A, Berardi N, Boldrini A, Cioni G, Maffei L. Massage accelerates brain development and the maturation of visual function. J Neurosci. 2009 May 6;29(18):6042-51. doi: 10.1523/JNEUROSCI.5548-08.2009. PMID 19420271
- [Background] Huguet G, Benabou M, Bourgeron T. The Genetics of Autism Spectrum Disorders. 2016 Apr 5. In: Sassone-Corsi P, Christen Y, editors. A Time for Metabolism and Hormones [Internet]. Cham (CH): Springer; 2016. Available from http://www.ncbi.nlm.nih.gov/books/NBK453174/ PMID 28892342
- [Background] Kong X, Liu J, Chien T, Batalden M, Hirsh DA. A Systematic Network of Autism Primary Care Services (SYNAPSE): A Model of Coproduction for the Management of Autism Spectrum Disorder. J Autism Dev Disord. 2020 May;50(5):1847-1853. doi: 10.1007/s10803-019-03922-4. PMID 30790194
- [Background] Lord C, Brugha TS, Charman T, Cusack J, Dumas G, Frazier T, Jones EJH, Jones RM, Pickles A, State MW, Taylor JL, Veenstra-VanderWeele J. Autism spectrum disorder. Nat Rev Dis Primers. 2020 Jan 16;6(1):5. doi: 10.1038/s41572-019-0138-4. PMID 31949163
- [Background] Luyster RJ, Wagner JB, Vogel-Farley V, Tager-Flusberg H, Nelson CA 3rd. Neural correlates of familiar and unfamiliar face processing in infants at risk for autism spectrum disorders. Brain Topogr. 2011 Oct;24(3-4):220-8. doi: 10.1007/s10548-011-0176-z. Epub 2011 Mar 26. PMID 21442325
- [Background] Maenner MJ, Warren Z, Williams AR, Amoakohene E, Bakian AV, Bilder DA, Durkin MS, Fitzgerald RT, Furnier SM, Hughes MM, Ladd-Acosta CM, McArthur D, Pas ET, Salinas A, Vehorn A, Williams S, Esler A, Grzybowski A, Hall-Lande J, Nguyen RHN, Pierce K, Zahorodny W, Hudson A, Hallas L, Mancilla KC, Patrick M, Shenouda J, Sidwell K, DiRienzo M, Gutierrez J, Spivey MH, Lopez M, Pettygrove S, Schwenk YD, Washington A, Shaw KA. Prevalence and Characteristics of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2020. MMWR Surveill Summ. 2023 Mar 24;72(2):1-14. doi: 10.15585/mmwr.ss7202a1. PMID 36952288
- [Background] Rutherford MD, Walsh JA, Lee V. Brief Report: Infants Developing with ASD Show a Unique Developmental Pattern of Facial Feature Scanning. J Autism Dev Disord. 2015 Aug;45(8):2618-23. doi: 10.1007/s10803-015-2396-7. PMID 25703032
- [Background] Saresella M, Marventano I, Guerini FR, Mancuso R, Ceresa L, Zanzottera M, Rusconi B, Maggioni E, Tinelli C, Clerici M. An autistic endophenotype results in complex immune dysfunction in healthy siblings of autistic children. Biol Psychiatry. 2009 Nov 15;66(10):978-84. doi: 10.1016/j.biopsych.2009.06.020. Epub 2009 Aug 22. PMID 19699471
- [Background] Wade L, Needham L, McGuigan P, Bilzon J. Applications and limitations of current markerless motion capture methods for clinical gait biomechanics. PeerJ. 2022 Feb 25;10:e12995. doi: 10.7717/peerj.12995. eCollection 2022. PMID 35237469
- [Background] Whittingham K, McGlade A, Kulasinghe K, Mitchell AE, Heussler H, Boyd RN. ENACT (ENvironmental enrichment for infants; parenting with Acceptance and Commitment Therapy): a randomised controlled trial of an innovative intervention for infants at risk of autism spectrum disorder. BMJ Open. 2020 Aug 20;10(8):e034315. doi: 10.1136/bmjopen-2019-034315. PMID 32819928
- [Derived] Annunziata S, Purpura G, Piazza E, Meriggi P, Fassina G, Santos L, Ambrosini E, Marchetti A, Manzi F, Massaro D, Tacci AL, Bolognesi E, Agostini S, La Rosa F, Pedrocchi APG, Molina P, Cavallini A. Early Recognition and Intervention in SIBlingS at High Risk for Neurodevelopment Disorders (ERI-SIBS): a controlled trial of an innovative and ecological intervention for siblings of children with autism spectrum disorder. Front Pediatr. 2025 Jan 6;12:1467783. doi: 10.3389/fped.2024.1467783. eCollection 2024. PMID 39834490